CLINICAL TRIAL: NCT00826553
Title: Comparison of Polysomnographic Findings in Mechanically Ventilated Patients Sedated With α2 Agonists Versus GABA Agonists
Brief Title: How Your Patients' Non-REM Sleep Changes On Sedatives in the Intensive Care Units
Acronym: HYPNOS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Wes Ely, Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 081170
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Delirium; Respiratory Failure
Keywords: sedative; GABA; alpha 2 agonist; propofol; midazolam; lorazepam; dexmedetomidine; sleep; electroencephalogram; polysomnogram; ICU
MeSH Terms: conditions — Delirium; Respiratory Insufficiency | interventions — Dexmedetomidine; GABA Agonists; Propofol; Midazolam; Lorazepam

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GABA agonist (Experimental)
  Interventions: Drug: GABA agonist
- Alpha 2 agonist (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Standard of care sedative. Dosage, frequency, and duration will be determined by the managing clinical team.
  Arms: Alpha 2 agonist
Drug: GABA agonist — Patients sedated with GABA agonists (e.g. propofol, benzodiazepines) during mechanical ventilation will be enrolled. Patients randomized to the GABA agonist arm will continue the sedative that is active at enrollment. The specific drug as well as dosage, frequency, and duration will be determined and titrated by the managing clinical team.
  Other Names: Typical GABA agonists include:; 1) propofol; 2) midazolam; 3) lorazepam.
  Arms: GABA agonist

SUMMARY:
The purpose of this study is to study the effect of two standard of care sedative medications on sleep stages and total sleep time. The investigators hypothesize that the α2 agonist, dexmedetomidine, will improve sleep quality by increasing N2 and N3 sleep as well as total sleep time when compared to GABA agonists.

DETAILED DESCRIPTION:
This is a single center randomized pilot study comparing the effects of an α2 agonist (dexmedetomidine) versus GABA agonists (propofol or a benzodiazepine) on total sleep time and sleep quality. For the purposes of enrollment and analysis all benzodiazepines used for sedation (mainly midazolam and lorazepam) will be considered equivalent. Patients who are mechanically ventilated and sedated will be enrolled. The initial sedative will be determined by the managing medical team and the medication will be active at the time of enrollment. The patients will then be randomized to either continue their current sedative or be switched to either propofol or dexmedetomidine. PSG data will be collected for up to 96 hours, beginning at enrollment for all patients. The analysis of PSG will not begin until after a 8 hour "washout" period has completed to minimize carryover effect of prior sedatives.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the medical intensive care unit who require mechanical ventilation and are sedated with a GABA agonist with the expectation of being mechanically ventilated for greater than 24 hours.

Exclusion Criteria:

* Subjects who are less than 18 years
* Subjects who are pregnant (a pregnancy test will be performed on all women of child bearing age)
* Inability to obtain informed consent from the patient or his/her surrogate
* Subjects who are physiologically benzodiazepine dependent, and at risk of withdrawal syndromes
* Subjects with anoxic brain injuries, strokes, or neurotrauma
* Medical team following patient unwilling to change sedation regimen
* Subjects who are moribund and not expected to survive 24 hours or actively withdrawing medical support
* Documented allergy to study medications
* Subjects with advanced heart block at time of screening
* Prisoners
* RASS target of less than or equal to -4 at the time of screening
* PSG equipment unavailable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Time spent in standard sleep stages (N1, N2, N3, REM). | 4 days

SECONDARY OUTCOMES:
Time spent in atypical sleep. | 4 days
Presence of burst suppression. | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Paula L Watson, MD, Principal Investigator — Vanderbilt School of Medicine
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States